CLINICAL TRIAL: NCT04977323
Title: Comparing The Effectiveness of Tracing Image and Coloring for Kids-Book With Two Passive Distractions on Pain and Fear in Children During Peripheral Intravenous Cannulation: A Randomized Controlled Trial
Brief Title: Comparison Effectiveness of Distractions on Pain and Fear of Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Principal Investigator, Sherzad Khudeida Suleman, Principal Investigator (PhD Student), University of Witten/Herdecke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Sherzad
Record Dates: First submitted 2021-07-04; First posted 2021-07-26 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Peripheral Intravenous Cannulation
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TICK-B group as intervention group (Experimental): TICK-B group: The children will receive the pictures they want. They will be asked to trace and color the pictures that need coloring. The nurse will color with children during the procedure. And after the procedure, the child will take his or her picture which he colored during the procedure.
  Interventions: Other: TICK-B group
- Watching cartoons (Experimental): Watching cartoons: In this group, children will watch cartoons as they like. Watching will continue until the procedure is complete.
  Interventions: Other: TICK-B group
- Group listening to music (Experimental): Listening to music: In this group, children will listen to cartoon music as they like. Listen will continue until the procedure is complete.
  Interventions: Other: TICK-B group
- Standard care provided group as control group (No Intervention): Control group. The kids in this group will be allowed to keep their family near. The routine blood taking

INTERVENTIONS:
Other: TICK-B group — These interventions will use as distraction techniques.
  Other Names: Watching cartoons; Listening to music group; Control group or no intervention
  Arms: Group listening to music; TICK-B group as intervention group; Watching cartoons

SUMMARY:
Distraction is a non-pharmacological technique that moves focus away from anxiety, discomfort or unpleasant stimulation to more stimulating or friendly stimulation. Distraction is one of the most effective, simplest and inexpensive non-pharmacological pain management methods (Hockenberry & Wilson, 2018). The benefits of using non-pharmacological methods include decreased pain, distress, and fear reported by the parent, child, and/or observer (Wente, 2013). There are two main types of distraction techniques: active and passive (Mutlu & Balcı, 2015; Wohlheiter & Dahlquist, 2013).

Objectives:

To evaluate the roles of the TICK-B, listening music, and watching cartoon, in relieving pain and fear of school-age children during PIVC.

To compare the effect of TICK-B with the effects of the listening music, and watching cartoon, on reducing pain and fear during PIVC in children.

To compare the effects of three distraction groups with the control group in relieving pain and fear during PIVC.

DETAILED DESCRIPTION:
Peripheral intravenous cannulation (PIVC) is an invasive technique. In this technique, a catheter is entrenched through the skin of the recipient into the lumen of a peripheral blood vein. It is the second most painful procedure performed in hospitals. Peripheral intravenous cannulation (PICV) is a common painful procedure for children, and nearly all ill children have experience with PIVC, and up to 80% of patients receive a peripheral venous cannula in a hospital. Therefore, the use of effective methods in pain and anxiety relief is very important during injection procedures in children.

In order to relieve pain and fear in children undergoing PICV. Psychological and physical approaches for coping with children's pain are favored, as well as pharmacological methods. Application of topical anesthetic creams is the most commonly used pharmacological solution to reduce pain associated with the medical procedure, or refrigerant preparations, however, only reduce the perception of pain in children during procedures. These approaches are not resolved anxiety, a core factor of noncooperation, which encumbers the efficiency of the needle procedure. For this cause, non-pharmacological approaches are generally recognized as alternative techniques, which may be used separately or in addition to pharmacological approaches, to provide sufficient pain and fear relief and to offer children a sense of control over the situation.

ELIGIBILITY:
Inclusion Criteria:

* School-aged 6-12 years old.
* Children who require PIVC.

Exclusion Criteria:

1. Respiratory chronic diseases,
2. Physical impairment,
3. Disability contributing to difficult communication,
4. Children of unsatisfied parents,
5. Children with neurodevelopment delay,
6. Cognitive impairment, hearing impairment or a visual impairment,
7. Taking an analgesic within 6 hours, or for those with a syncope history.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2021-07-28 (Estimated); Primary Completion 2021-10-05 (Estimated); Study Completion 2021-10-10 (Estimated)

PRIMARY OUTCOMES:
Faces Pain Scale-Revised to rate the severity of Pain (0-10) from no pain to worst pain | 5 minutes before procedure done.
  To assess the intensity of pain related to Peripheral intravenous cannulation procedure in children:
  Children will self-report their pain severity using the Faces Pain Scale-Revised, which has been validated and shown to be reliable.
Children's Fear Scale (CFS): Fear (0-4) no anxiety to extreme anxiety | 5 minutes before procedure done
  To assess the fear level of the children related to Peripheral intravenous cannulation procedure:
  Children will self-report their level of fear using the Children's Fear Scale (CFS), which has been validated and shown to be reliable.

SECONDARY OUTCOMES:
Faces Pain Scale-Revised to rate the severity of Pain (0-10) from no pain to worst pain. | 0 minute during peripheral cannulation insertion procedure(time during insertion of cannula).
  To assess the intensity of pain related to Peripheral intravenous cannulation procedure in children:
  Children will self-report their pain severity using the Faces Pain Scale-Revised, which has been validated and shown to be reliable.
Faces Pain Scale-Revised to rate the severity of Pain (0-10) from no pain to worst pain. | 1-2 minutes after procedure done.
  To assess the intensity of pain related to peripheral intravenous cannulation procedure in children:
  Children will self-report their pain severity using the Faces Pain Scale-Revised, which has been validated and shown to be reliable.
Children's Fear Scale (CFS): Fear (0-4) no anxiety to extreme anxiety | 0 minute during cannulation procedure.
  To assess the fear level of the children related to peripheral intravenous cannulation procedure:
  -Children will self-report their level of fear using the Children's Fear Scale (CFS), which has been validated and shown to be reliable.
Children's Fear Scale (CFS): Fear (0-4) no anxiety to extreme anxiety | 1-2 minute after cannulation procedure done.
  To assess the fear level of the children related to peripheral intravenous cannulation procedure:
  -Children will self-report their level of fear using the Children's Fear Scale (CFS), which has been validated and shown to be reliable.

OTHER OUTCOMES:
Visual Analog Scale (VAS), to measure the pain and Fear of children by the parents and observer. | Immediately after cannualtion (1-2 minutes after procedure to mask observer)
  Visual Analog Scale (VAS) will be used to measure pain and fear of children by parent and observer.

REFERENCES:
- [Background] Hockenberry, M. J., & Wilson, D. (2018). Wong's nursing care of infants and children-E-book. Elsevier Health Sciences.
- [Background] Wente SJ. Nonpharmacologic pediatric pain management in emergency departments: a systematic review of the literature. J Emerg Nurs. 2013 Mar;39(2):140-50. doi: 10.1016/j.jen.2012.09.011. Epub 2012 Nov 28. PMID 23199786
- [Background] Mutlu B, Balci S. Effects of balloon inflation and cough trick methods on easing pain in children during the drawing of venous blood samples: a randomized controlled trial. J Spec Pediatr Nurs. 2015 Jul;20(3):178-86. doi: 10.1111/jspn.12112. Epub 2015 Mar 28. PMID 25817062
- [Background] Hendry F, Checketts MR, McLeod GA. Effect of intradermal anaesthesia on success rate and pain of intravenous cannulation: a randomized non-blind crossover study. Scott Med J. 2011 Nov;56(4):210-3. doi: 10.1258/smj.2011.011160. PMID 22089042
- [Background] Rogers TL, Ostrow CL. The use of EMLA cream to decrease venipuncture pain in children. J Pediatr Nurs. 2004 Feb;19(1):33-9. doi: 10.1016/j.pedn.2003.09.005. PMID 14963868
- [Background] Blount RL, Piira T, Cohen LL, Cheng PS. Pediatric procedural pain. Behav Modif. 2006 Jan;30(1):24-49. doi: 10.1177/0145445505282438. PMID 16330518
- [Background] Friedrichsdorf SJ, Eull D, Weidner C, Postier A. A hospital-wide initiative to eliminate or reduce needle pain in children using lean methodology. Pain Rep. 2018 Sep 11;3(Suppl 1):e671. doi: 10.1097/PR9.0000000000000671. eCollection 2018 Sep. PMID 30324169
- [Background] Shomaker K, Dutton S, Mark M. Pain Prevalence and Treatment Patterns in a US Children's Hospital. Hosp Pediatr. 2015 Jul;5(7):363-70. doi: 10.1542/hpeds.2014-0195. PMID 26136310
- [Background] Uman LS, Chambers CT, McGrath PJ, Kisely S. A systematic review of randomized controlled trials examining psychological interventions for needle-related procedural pain and distress in children and adolescents: an abbreviated cochrane review. J Pediatr Psychol. 2008 Sep;33(8):842-54. doi: 10.1093/jpepsy/jsn031. Epub 2008 Apr 2. PMID 18387963